CLINICAL TRIAL: NCT05333679
Title: Urine Tenofovir Point-of-care Test to Identify Patients in Need of ART Adherence Support (UTRA Study)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Cape Town (Other); University of Stellenbosch (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AI152119; 5R01AI152119 (NIH)
Record Dates: First submitted 2022-04-11; First posted 2022-04-19 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Risk Reduction
Keywords: UTRA; Point-of-care; Real-time; PLHIV; Adherence monitoring; ART
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intervention (Experimental): POC adherence testing by a urine TFV assay with feedback
  Interventions: Device: UTRA; Behavioral: UTRA feedback
- Standard of Care (No Intervention): Standard enhanced adherence counselling, SA Department of Health, March 2020

INTERVENTIONS:
Device: UTRA — Collect urine on intervention participants and screen for presence of TFV.
  Arms: Intervention
Behavioral: UTRA feedback — Feedback will be provided to the participant based on the UTRA results on their adherence with provision of standard adherence counseling.
  Arms: Intervention

SUMMARY:
ART is given to people living with HIV in order to suppress the virus, resulting in improved health for the individual and decreased transmission of the virus to others. Success of ART is dependent on adherence. Currently, adherence is assessed by asking patients directly and then confirming with a viral load test, which is expensive and is often only done when the viral load is already raised. Therefore there is a need to find a method to detect problems with adherence early before the viral load rises.

A urine-based test was recently developed, called UTRA (urine tenofovir rapid assay). This test can give clinic staff immediate results about a person's adherence to the antiretroviral medication Tenofovir (TDF). The study will compare the results of this urine test to drug levels found in blood, self-reported adherence and pharmacy collection records to see if this test can be used as part of routine care in ART clinics. If the test is effective it would allow clinic staff to identify people with adherence difficulties early and give them the necessary support before their viral load rises.

DETAILED DESCRIPTION:
This is a randomised study, recruiting 200 people taking TDF-based ART. Participants will be randomised 1:1 to intervention versus standard enhanced adherence counselling. Intervention participants will receive an adherence support package informed by feedback from the urine-based test. The investigators will assess the impact of the adherence test on VL suppression rates in each arm (without necessitating a regimen switch) at 12 months after enrolment. Enrolling participants with adherence challenges increases efficiency and mirrors the population requiring adherence support in our setting.

The UTRA device used for this study has received a FDA Non-Significant Risk (NSR) designation and is IDE exempt.

FEASIBILITY:

The investigators will track retention in the study among participants in each arm, missed visits, and the number of urine assessments performed in the intervention arm.

ACCEPTABILITY:

All participants enrolled will also complete a standardised questionnaire about the acceptability of the adherence support they received. This measure of acceptability will be assessed as a secondary outcome by arm, along with socio-demographics profiles associated with low/high acceptability described within arm.

QUALITATIVE PROCEDURES:

1. Participant in-depth interviews: Qualitative data will include in-depth interviews of participants (n~20; ~3-4 interviews with each participant over 6-9 months of their treatment) using semi-structured guides conducted by experienced socio-behavioural scientists. The semi-structured interview guide will elicit feelings about the urine adherence metric and counseling messages, concerns regarding privacy, advantages/disadvantages of receiving such results, and the likely impact of this monitoring test on sustained adherence to ART or just on short-term adherence. Interviews will be conducted in participants' preferred language.
2. Health care worker interviews: The investigators will additionally assess the feasibility of the intervention by interviewing health care providers, who will be administering the UTRA test at the clinical point of care in the future. The study will examine provider perceptions of the assay at the end of the study using in-depth interviews (n~10), assessing perceived usefulness, complexity to use, stigma/social harm, and benefits. These interviews will also elicit barriers and facilitators to delivery of the urine assay-informed counseling messages.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Willing and able to provide written informed consent
* HIV-infected, receiving or (re-)starting a tenofovir-based ART regimen
* Current ART regimen includes at least one drug with a high genetic barrier to resistance e.g. dolutegravir, atazanavir/ritonavir, darunavir/ritonavir or lopinavir/ritonavir.
* Any previous raised viral load >50 copies/ml (after ART initiation).
* Willing and able to comply with laboratory tests and other study procedures

Exclusion Criteria:

* Not willing or able to provide informed consent in any of the languages provided
* Not receiving a tenofovir-based ART regimen
* Any other clinical condition that in the opinion of an investigator puts the patient at increased risk if participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants in each arm achieving viral suppression to <50 copies/ml | 21 months
  Assess suppression rates (VL< 50 copies/mL) in both study arms using an intention-to-treat analysis. Plasma will be stored an enrolment, month 6 and month 12 for viral load assay completion after the study. Samples are assayed either with the Alinity m HIV-1 assay (Abbott Laboratories. Abbott Park, Illinois, U.S.A.); lower limit of detection (LLD) 10 copies/mL or the COBAS® AmpliPrep/COBAS® TaqMan® HIV-1 Test, v2.0 (Roche Diagnostics, Basel, Switzerland); LLD 20 copies/mL. Whole blood will be centrifuged and plasma then tested on the automated analyzer according to national standard operating procedures

SECONDARY OUTCOMES:
Retention in care | 21 months
  Follow up visits will occur in 12-week increments post-enrolment: at month 3, month 6, month 9 and month 12; and will be synchronized wherever possible with routine clinic visits. Visit windows will be continuous, with each window extending to 6 weeks before and 6 weeks after the visit target date. A visit will be considered missed if the participant does not attend during the 12-week visit window
Viral suppression (<50 copies/mL) | 21 months
  Assess suppression rates (VL< 50 copies/mL) in both study arms using an intention-to-treat analysis. Samples are assayed either with the Alinity m HIV-1 assay (Abbott Laboratories. Abbott Park, Illinois, U.S.A.); lower limit of detection (LLD) 10 copies/mL or the COBAS® AmpliPrep/COBAS® TaqMan® HIV-1 Test, v2.0 (Roche Diagnostics, Basel, Switzerland); LLD 20 copies/mL. Whole blood will be centrifuged and plasma then tested on the automated analyzer according to national standard operating procedures
The proportion of participants indicating "strongly agree" or "agree" averaged across 10 items, each using a five-point Likert scale to measure aspects of the adherence support intervention (i.e., by arm: UTRA-informed or standard of care) | 21 months
  The proportion of participants indicating "strongly agree" or "agree" averaged across 10 items, each item using a five-point Likert scale to measure aspects of acceptability of the adherence support intervention (i.e., by arm: UTRA-informed or standard of care), at month 12. Responses to the Likert scale range from "Strongly agree" to "Strongly disagree". Aspects of acceptability include domains on: support from health workers, time given by health workers to discuss the patients' treatment, patient perceptions of feeling informed about their adherence, feelings of surveillance (-vely scored), and self-satisfactions with adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Gandhi, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Desmond Tutu Health Foundation, University of Cape Town, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Yes
We will share de-identified data in publicly accessible databases once study is complete and study findings disseminated.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 48 months from start of study
Access Criteria: Investigators conducting PrEP research

REFERENCES:
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Cottle L, Zhang XC, Makhema J, Mills LA, Panchia R, Faesen S, Eron J, Gallant J, Havlir D, Swindells S, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano DD, Essex M, Hudelson SE, Redd AD, Fleming TR; HPTN 052 Study Team. Antiretroviral Therapy for the Prevention of HIV-1 Transmission. N Engl J Med. 2016 Sep 1;375(9):830-9. doi: 10.1056/NEJMoa1600693. Epub 2016 Jul 18. PMID 27424812
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Mehendale S, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Wang L, Makhema J, Mills LA, de Bruyn G, Sanne I, Eron J, Gallant J, Havlir D, Swindells S, Ribaudo H, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano D, Essex M, Fleming TR; HPTN 052 Study Team. Prevention of HIV-1 infection with early antiretroviral therapy. N Engl J Med. 2011 Aug 11;365(6):493-505. doi: 10.1056/NEJMoa1105243. Epub 2011 Jul 18. PMID 21767103
- [Background] Rodger AJ, Cambiano V, Bruun T, Vernazza P, Collins S, Degen O, Corbelli GM, Estrada V, Geretti AM, Beloukas A, Raben D, Coll P, Antinori A, Nwokolo N, Rieger A, Prins JM, Blaxhult A, Weber R, Van Eeden A, Brockmeyer NH, Clarke A, Del Romero Guerrero J, Raffi F, Bogner JR, Wandeler G, Gerstoft J, Gutierrez F, Brinkman K, Kitchen M, Ostergaard L, Leon A, Ristola M, Jessen H, Stellbrink HJ, Phillips AN, Lundgren J; PARTNER Study Group. Risk of HIV transmission through condomless sex in serodifferent gay couples with the HIV-positive partner taking suppressive antiretroviral therapy (PARTNER): final results of a multicentre, prospective, observational study. Lancet. 2019 Jun 15;393(10189):2428-2438. doi: 10.1016/S0140-6736(19)30418-0. Epub 2019 May 2. PMID 31056293
- [Background] Rodger AJ, Cambiano V, Bruun T, Vernazza P, Collins S, van Lunzen J, Corbelli GM, Estrada V, Geretti AM, Beloukas A, Asboe D, Viciana P, Gutierrez F, Clotet B, Pradier C, Gerstoft J, Weber R, Westling K, Wandeler G, Prins JM, Rieger A, Stoeckle M, Kummerle T, Bini T, Ammassari A, Gilson R, Krznaric I, Ristola M, Zangerle R, Handberg P, Antela A, Allan S, Phillips AN, Lundgren J; PARTNER Study Group. Sexual Activity Without Condoms and Risk of HIV Transmission in Serodifferent Couples When the HIV-Positive Partner Is Using Suppressive Antiretroviral Therapy. JAMA. 2016 Jul 12;316(2):171-81. doi: 10.1001/jama.2016.5148. PMID 27404185
- [Background] Herzer M, Ramey C, Rohan J, Cortina S. Incorporating electronic monitoring feedback into clinical care: a novel and promising adherence promotion approach. Clin Child Psychol Psychiatry. 2012 Oct;17(4):505-18. doi: 10.1177/1359104511421103. Epub 2011 Sep 25. PMID 21949048
- [Background] de Necker M, de Beer JC, Stander MP, Connell CD, Mwai D. Economic and public health impact of decentralized HIV viral load testing: A modelling study in Kenya. PLoS One. 2019 Feb 27;14(2):e0212972. doi: 10.1371/journal.pone.0212972. eCollection 2019. PMID 30811510
- [Background] van Zyl GU, van Mens TE, McIlleron H, Zeier M, Nachega JB, Decloedt E, Malavazzi C, Smith P, Huang Y, van der Merwe L, Gandhi M, Maartens G. Low lopinavir plasma or hair concentrations explain second-line protease inhibitor failures in a resource-limited setting. J Acquir Immune Defic Syndr. 2011 Apr;56(4):333-9. doi: 10.1097/QAI.0b013e31820dc0cc. PMID 21239995
- [Background] Prasitsuebsai W, Kerr SJ, Truong KH, Ananworanich J, Do VC, Nguyen LV, Kurniati N, Kosalaraksa P, Sudjaritruk T, Chokephaibulkit K, Thammajaruk N, Singtoroj T, Teeraananchai S, Horng H, Bacchetti P, Gandhi M, Sohn AH. Using Lopinavir Concentrations in Hair Samples to Assess Treatment Outcomes on Second-Line Regimens Among Asian Children. AIDS Res Hum Retroviruses. 2015 Oct;31(10):1009-14. doi: 10.1089/AID.2015.0111. Epub 2015 Aug 26. PMID 26200586
- [Background] Murnane PM, Bacchetti P, Currier JS, Brummel S, Okochi H, Phung N, Louie A, Kuncze K, Hoffman RM, Nematadzira T, Soko DK, Owor M, Saidi F, Flynn PM, Fowler MG, Gandhi M. Tenofovir concentrations in hair strongly predict virologic suppression in breastfeeding women. AIDS. 2019 Aug 1;33(10):1657-1662. doi: 10.1097/QAD.0000000000002237. PMID 31021852
- [Background] Gandhi M, Bacchetti P, Ofokotun I, Jin C, Ribaudo HJ, Haas DW, Sheth AN, Horng H, Phung N, Kuncze K, Okochi H, Landovitz RJ, Lennox J, Currier JS; AIDS Clinical Trials Group (ACTG) 5257 Study Team. Antiretroviral Concentrations in Hair Strongly Predict Virologic Response in a Large Human Immunodeficiency Virus Treatment-naive Clinical Trial. Clin Infect Dis. 2019 Mar 5;68(6):1044-1047. doi: 10.1093/cid/ciy764. PMID 30184104
- [Background] Gandhi M, Ameli N, Bacchetti P, Gange SJ, Anastos K, Levine A, Hyman CL, Cohen M, Young M, Huang Y, Greenblatt RM; Women's Interagency HIV Study (WIHS). Protease inhibitor levels in hair strongly predict virologic response to treatment. AIDS. 2009 Feb 20;23(4):471-8. doi: 10.1097/QAD.0b013e328325a4a9. PMID 19165084
- [Background] Gandhi M, Ameli N, Bacchetti P, Anastos K, Gange SJ, Minkoff H, Young M, Milam J, Cohen MH, Sharp GB, Huang Y, Greenblatt RM. Atazanavir concentration in hair is the strongest predictor of outcomes on antiretroviral therapy. Clin Infect Dis. 2011 May;52(10):1267-75. doi: 10.1093/cid/cir131. PMID 21507924
- [Background] Cohan D, Natureeba P, Koss CA, Plenty A, Luwedde F, Mwesigwa J, Ades V, Charlebois ED, Gandhi M, Clark TD, Nzarubara B, Achan J, Ruel T, Kamya MR, Havlir DV. Efficacy and safety of lopinavir/ritonavir versus efavirenz-based antiretroviral therapy in HIV-infected pregnant Ugandan women. AIDS. 2015 Jan 14;29(2):183-91. doi: 10.1097/QAD.0000000000000531. PMID 25426808
- [Background] Koss CA, Natureeba P, Mwesigwa J, Cohan D, Nzarubara B, Bacchetti P, Horng H, Clark TD, Plenty A, Ruel TD, Achan J, Charlebois ED, Kamya MR, Havlir DV, Gandhi M. Hair concentrations of antiretrovirals predict viral suppression in HIV-infected pregnant and breastfeeding Ugandan women. AIDS. 2015 Apr 24;29(7):825-30. doi: 10.1097/QAD.0000000000000619. PMID 25985404
- [Background] Chawana TD, Gandhi M, Nathoo K, Ngara B, Louie A, Horng H, Katzenstein D, Metcalfe J, Nhachi CFB; Adolescent Treatment Failure (ATF) study team. Defining a Cutoff for Atazanavir in Hair Samples Associated With Virological Failure Among Adolescents Failing Second-Line Antiretroviral Treatment. J Acquir Immune Defic Syndr. 2017 Sep 1;76(1):55-59. doi: 10.1097/QAI.0000000000001452. PMID 28520618
- [Background] Pintye J, Bacchetti P, Teeraananchai S, Kerr S, Prasitsuebsai W, Singtoroj T, Kuncze K, Louie A, Koss CA, Jin C, Phung N, Horng H, Sohn AH, Gandhi M. Brief Report: Lopinavir Hair Concentrations Are the Strongest Predictor of Viremia in HIV-Infected Asian Children and Adolescents on Second-Line Antiretroviral Therapy. J Acquir Immune Defic Syndr. 2017 Dec 1;76(4):367-371. doi: 10.1097/QAI.0000000000001527. PMID 28825944
- [Background] Baxi SM, Greenblatt RM, Bacchetti P, Jin C, French AL, Keller MJ, Augenbraun MH, Gange SJ, Liu C, Mack WJ, Gandhi M; Women's Interagency HIV Study (WIHS). Nevirapine Concentration in Hair Samples Is a Strong Predictor of Virologic Suppression in a Prospective Cohort of HIV-Infected Patients. PLoS One. 2015 Jun 8;10(6):e0129100. doi: 10.1371/journal.pone.0129100. eCollection 2015. PMID 26053176
- [Background] Tabb ZJ, Mmbaga BT, Gandhi M, Louie A, Kuncze K, Okochi H, Shayo AM, Turner EL, Cunningham CK, Dow DE. Antiretroviral drug concentrations in hair are associated with virologic outcomes among young people living with HIV in Tanzania. AIDS. 2018 Jun 1;32(9):1115-1123. doi: 10.1097/QAD.0000000000001788. PMID 29438196
- [Background] Marrazzo JM, Ramjee G, Richardson BA, Gomez K, Mgodi N, Nair G, Palanee T, Nakabiito C, van der Straten A, Noguchi L, Hendrix CW, Dai JY, Ganesh S, Mkhize B, Taljaard M, Parikh UM, Piper J, Masse B, Grossman C, Rooney J, Schwartz JL, Watts H, Marzinke MA, Hillier SL, McGowan IM, Chirenje ZM; VOICE Study Team. Tenofovir-based preexposure prophylaxis for HIV infection among African women. N Engl J Med. 2015 Feb 5;372(6):509-18. doi: 10.1056/NEJMoa1402269. PMID 25651245
- [Background] Gandhi M, Bacchetti P, Rodrigues WC, Spinelli M, Koss CA, Drain PK, Baeten JM, Mugo NR, Ngure K, Benet LZ, Okochi H, Wang G, Vincent M. Development and Validation of an Immunoassay for Tenofovir in Urine as a Real-Time Metric of Antiretroviral Adherence. EClinicalMedicine. 2018 Aug-Sep;2-3:22-28. doi: 10.1016/j.eclinm.2018.08.004. Epub 2018 Aug 31. PMID 30906930
- [Background] Castillo-Mancilla JR, Zheng JH, Rower JE, Meditz A, Gardner EM, Predhomme J, Fernandez C, Langness J, Kiser JJ, Bushman LR, Anderson PL. Tenofovir, emtricitabine, and tenofovir diphosphate in dried blood spots for determining recent and cumulative drug exposure. AIDS Res Hum Retroviruses. 2013 Feb;29(2):384-90. doi: 10.1089/AID.2012.0089. Epub 2012 Oct 10. PMID 22935078
- [Background] Gandhi M, Greenblatt RM. Hair it is: the long and short of monitoring antiretroviral treatment. Ann Intern Med. 2002 Oct 15;137(8):696-7. doi: 10.7326/0003-4819-137-8-200210150-00016. No abstract available. PMID 12379072
- [Background] DePriest AZ, Black DL, Robert TA. Immunoassay in healthcare testing applications. J Opioid Manag. 2015 Jan-Feb;11(1):13-25. doi: 10.5055/jom.2015.0248. PMID 25750161
- [Background] Pecoraro V, Banfi G, Germagnoli L, Trenti T. A systematic evaluation of immunoassay point-of-care testing to define impact on patients' outcomes. Ann Clin Biochem. 2017 Jul;54(4):420-431. doi: 10.1177/0004563217694377. Epub 2017 May 15. PMID 28135840
- [Background] Zash R, Makhema J, Shapiro RL. Neural-Tube Defects with Dolutegravir Treatment from the Time of Conception. N Engl J Med. 2018 Sep 6;379(10):979-981. doi: 10.1056/NEJMc1807653. Epub 2018 Jul 24. No abstract available. PMID 30037297
- [Background] Keene CM, Griesel R, Zhao Y, Gcwabe Z, Sayed K, Hill A, Cassidy T, Ngwenya O, Jackson A, van Zyl G, Schutz C, Goliath R, Flowers T, Goemaere E, Wiesner L, Simmons B, Maartens G, Meintjes G. Virologic efficacy of tenofovir, lamivudine and dolutegravir as second-line antiretroviral therapy in adults failing a tenofovir-based first-line regimen. AIDS. 2021 Jul 15;35(9):1423-1432. doi: 10.1097/QAD.0000000000002936. PMID 33973876
- [Background] Gandhi M, Bacchetti P, Spinelli MA, Okochi H, Baeten JM, Siriprakaisil O, Klinbuayaem V, Rodrigues WC, Wang G, Vincent M, Cressey TR, Drain PK. Brief Report: Validation of a Urine Tenofovir Immunoassay for Adherence Monitoring to PrEP and ART and Establishing the Cutoff for a Point-of-Care Test. J Acquir Immune Defic Syndr. 2019 May 1;81(1):72-77. doi: 10.1097/QAI.0000000000001971. PMID 30664078
- [Background] Cressey TR, Siriprakaisil O, Klinbuayaem V, Quame-Amaglo J, Kubiak RW, Sukrakanchana PO, Than-In-At K, Baeten J, Sirirungsi W, Cressey R, Drain PK. A randomized clinical pharmacokinetic trial of Tenofovir in blood, plasma and urine in adults with perfect, moderate and low PrEP adherence: the TARGET study. BMC Infect Dis. 2017 Jul 14;17(1):496. doi: 10.1186/s12879-017-2593-4. PMID 28705153
- [Background] Koenig HC, Mounzer K, Daughtridge GW, Sloan CE, Lalley-Chareczko L, Moorthy GS, Conyngham SC, Zuppa AF, Montaner LJ, Tebas P. Urine assay for tenofovir to monitor adherence in real time to tenofovir disoproxil fumarate/emtricitabine as pre-exposure prophylaxis. HIV Med. 2017 Jul;18(6):412-418. doi: 10.1111/hiv.12518. Epub 2017 Apr 26. PMID 28444867
- [Background] Marrazzo JM, Scholes D. Acceptability of urine-based screening for Chlamydia trachomatis in asymptomatic young men: a systematic review. Sex Transm Dis. 2008 Nov;35(11 Suppl):S28-33. doi: 10.1097/OLQ.0b013e31816938ca. PMID 18418291
- [Background] Hadland SE, Levy S. Objective Testing: Urine and Other Drug Tests. Child Adolesc Psychiatr Clin N Am. 2016 Jul;25(3):549-65. doi: 10.1016/j.chc.2016.02.005. Epub 2016 Mar 30. PMID 27338974
- [Background] Spinelli MA, Glidden DV, Rodrigues WC, Wang G, Vincent M, Okochi H, Kuncze K, Mehrotra M, Defechereux P, Buchbinder SP, Grant RM, Gandhi M. Low tenofovir level in urine by a novel immunoassay is associated with seroconversion in a preexposure prophylaxis demonstration project. AIDS. 2019 Apr 1;33(5):867-872. doi: 10.1097/QAD.0000000000002135. PMID 30649051
- [Background] Parienti JJ, Das-Douglas M, Massari V, Guzman D, Deeks SG, Verdon R, Bangsberg DR. Not all missed doses are the same: sustained NNRTI treatment interruptions predict HIV rebound at low-to-moderate adherence levels. PLoS One. 2008 Jul 30;3(7):e2783. doi: 10.1371/journal.pone.0002783. PMID 18665246
- [Background] Parienti JJ, Ragland K, Lucht F, de la Blanchardiere A, Dargere S, Yazdanpanah Y, Dutheil JJ, Perre P, Verdon R, Bangsberg DR; ESPOIR and REACH study groups. Average adherence to boosted protease inhibitor therapy, rather than the pattern of missed doses, as a predictor of HIV RNA replication. Clin Infect Dis. 2010 Apr 15;50(8):1192-7. doi: 10.1086/651419. PMID 20210643
- [Background] Gandhi M, Glidden DV, Liu A, Anderson PL, Horng H, Defechereux P, Guanira JV, Grinsztejn B, Chariyalertsak S, Bekker LG, Grant RM; iPrEx Study Team. Strong Correlation Between Concentrations of Tenofovir (TFV) Emtricitabine (FTC) in Hair and TFV Diphosphate and FTC Triphosphate in Dried Blood Spots in the iPrEx Open Label Extension: Implications for Pre-exposure Prophylaxis Adherence Monitoring. J Infect Dis. 2015 Nov 1;212(9):1402-6. doi: 10.1093/infdis/jiv239. Epub 2015 Apr 20. PMID 25895984
- [Background] Gandhi M, Murnane PM, Bacchetti P, Elion R, Kolber MA, Cohen SE, Horng H, Louie A, Kuncze K, Koss CA, Anderson PL, Buchbinder S, Liu A. Hair levels of preexposure prophylaxis drugs measure adherence and are associated with renal decline among men/transwomen. AIDS. 2017 Oct 23;31(16):2245-2251. doi: 10.1097/QAD.0000000000001615. PMID 28832411
- [Background] Koss CA, Hosek SG, Bacchetti P, Anderson PL, Liu AY, Horng H, Benet LZ, Kuncze K, Louie A, Saberi P, Wilson CM, Gandhi M. Comparison of Measures of Adherence to Human Immunodeficiency Virus Preexposure Prophylaxis Among Adolescent and Young Men Who Have Sex With Men in the United States. Clin Infect Dis. 2018 Jan 6;66(2):213-219. doi: 10.1093/cid/cix755. PMID 29020194
- [Background] Van Damme L, Corneli A, Ahmed K, Agot K, Lombaard J, Kapiga S, Malahleha M, Owino F, Manongi R, Onyango J, Temu L, Monedi MC, Mak'Oketch P, Makanda M, Reblin I, Makatu SE, Saylor L, Kiernan H, Kirkendale S, Wong C, Grant R, Kashuba A, Nanda K, Mandala J, Fransen K, Deese J, Crucitti T, Mastro TD, Taylor D; FEM-PrEP Study Group. Preexposure prophylaxis for HIV infection among African women. N Engl J Med. 2012 Aug 2;367(5):411-22. doi: 10.1056/NEJMoa1202614. Epub 2012 Jul 11. PMID 22784040
- [Background] Grant RM, Lama JR, Anderson PL, McMahan V, Liu AY, Vargas L, Goicochea P, Casapia M, Guanira-Carranza JV, Ramirez-Cardich ME, Montoya-Herrera O, Fernandez T, Veloso VG, Buchbinder SP, Chariyalertsak S, Schechter M, Bekker LG, Mayer KH, Kallas EG, Amico KR, Mulligan K, Bushman LR, Hance RJ, Ganoza C, Defechereux P, Postle B, Wang F, McConnell JJ, Zheng JH, Lee J, Rooney JF, Jaffe HS, Martinez AI, Burns DN, Glidden DV; iPrEx Study Team. Preexposure chemoprophylaxis for HIV prevention in men who have sex with men. N Engl J Med. 2010 Dec 30;363(27):2587-99. doi: 10.1056/NEJMoa1011205. Epub 2010 Nov 23. PMID 21091279
- [Background] Van Damme L, Corneli A. Antiretroviral preexposure prophylaxis for HIV prevention. N Engl J Med. 2013 Jan 3;368(1):84. doi: 10.1056/NEJMc1210464. No abstract available. PMID 23293792
- [Background] Blumenthal J, Haubrich R. Pre-exposure prophylaxis for HIV infection: how antiretroviral pharmacology helps to monitor and improve adherence. Expert Opin Pharmacother. 2013 Sep;14(13):1777-85. doi: 10.1517/14656566.2013.812072. Epub 2013 Jun 26. PMID 23800167
- [Background] Musinguzi N, Muganzi CD, Boum Y 2nd, Ronald A, Marzinke MA, Hendrix CW, Celum C, Baeten JM, Bangsberg DR, Haberer JE; Partners PrEP Ancillary Adherence Study Team. Comparison of subjective and objective adherence measures for preexposure prophylaxis against HIV infection among serodiscordant couples in East Africa. AIDS. 2016 Apr 24;30(7):1121-9. doi: 10.1097/QAD.0000000000001024. PMID 26785125
- [Background] Donnell D, Baeten JM, Bumpus NN, Brantley J, Bangsberg DR, Haberer JE, Mujugira A, Mugo N, Ndase P, Hendrix C, Celum C. HIV protective efficacy and correlates of tenofovir blood concentrations in a clinical trial of PrEP for HIV prevention. J Acquir Immune Defic Syndr. 2014 Jul 1;66(3):340-8. doi: 10.1097/QAI.0000000000000172. PMID 24784763
- [Background] Thigpen MC, Kebaabetswe PM, Paxton LA, Smith DK, Rose CE, Segolodi TM, Henderson FL, Pathak SR, Soud FA, Chillag KL, Mutanhaurwa R, Chirwa LI, Kasonde M, Abebe D, Buliva E, Gvetadze RJ, Johnson S, Sukalac T, Thomas VT, Hart C, Johnson JA, Malotte CK, Hendrix CW, Brooks JT; TDF2 Study Group. Antiretroviral preexposure prophylaxis for heterosexual HIV transmission in Botswana. N Engl J Med. 2012 Aug 2;367(5):423-34. doi: 10.1056/NEJMoa1110711. Epub 2012 Jul 11. PMID 22784038
- [Background] Choopanya K, Martin M, Suntharasamai P, Sangkum U, Mock PA, Leethochawalit M, Chiamwongpaet S, Kitisin P, Natrujirote P, Kittimunkong S, Chuachoowong R, Gvetadze RJ, McNicholl JM, Paxton LA, Curlin ME, Hendrix CW, Vanichseni S; Bangkok Tenofovir Study Group. Antiretroviral prophylaxis for HIV infection in injecting drug users in Bangkok, Thailand (the Bangkok Tenofovir Study): a randomised, double-blind, placebo-controlled phase 3 trial. Lancet. 2013 Jun 15;381(9883):2083-90. doi: 10.1016/S0140-6736(13)61127-7. Epub 2013 Jun 13. PMID 23769234
- [Background] Haberer JE, Musinguzi N, Boum Y 2nd, Siedner MJ, Mocello AR, Hunt PW, Martin JN, Bangsberg DR. Duration of Antiretroviral Therapy Adherence Interruption Is Associated With Risk of Virologic Rebound as Determined by Real-Time Adherence Monitoring in Rural Uganda. J Acquir Immune Defic Syndr. 2015 Dec 1;70(4):386-92. doi: 10.1097/QAI.0000000000000737. PMID 26110445
- [Background] Steegen K, Bronze M, Papathanasopoulos MA, van Zyl G, Goedhals D, Variava E, MacLeod W, Sanne I, Stevens WS, Carmona S. HIV-1 antiretroviral drug resistance patterns in patients failing NNRTI-based treatment: results from a national survey in South Africa. J Antimicrob Chemother. 2017 Jan;72(1):210-219. doi: 10.1093/jac/dkw358. Epub 2016 Sep 22. PMID 27659733
- [Background] Orrell C, Walensky RP, Losina E, Pitt J, Freedberg KA, Wood R. HIV type-1 clade C resistance genotypes in treatment-naive patients and after first virological failure in a large community antiretroviral therapy programme. Antivir Ther. 2009;14(4):523-31. PMID 19578237
- [Background] Hoffmann CJ, Charalambous S, Sim J, Ledwaba J, Schwikkard G, Chaisson RE, Fielding KL, Churchyard GJ, Morris L, Grant AD. Viremia, resuppression, and time to resistance in human immunodeficiency virus (HIV) subtype C during first-line antiretroviral therapy in South Africa. Clin Infect Dis. 2009 Dec 15;49(12):1928-35. doi: 10.1086/648444. PMID 19911963
- [Background] Charpentier C, Peytavin G, Le MP, Joly V, Cabras O, Perrier M, Le Gac S, Phung B, Yazdanpanah Y, Descamps D, Landman R. High virological suppression regardless of the genotypic susceptibility score after switching to a dolutegravir-based regimen: week 48 results in an observational cohort. J Antimicrob Chemother. 2018 Jun 1;73(6):1665-1671. doi: 10.1093/jac/dky062. PMID 29528412
- [Background] Jacobson K, Ogbuagu O. Integrase inhibitor-based regimens result in more rapid virologic suppression rates among treatment-naive human immunodeficiency virus-infected patients compared to non-nucleoside and protease inhibitor-based regimens in a real-world clinical setting: A retrospective cohort study. Medicine (Baltimore). 2018 Oct;97(43):e13016. doi: 10.1097/MD.0000000000013016. PMID 30412140
- [Background] Rahangdale L, Cates J, Potter J, Badell ML, Seidman D, Miller ES, Coleman JS, Lazenby GB, Levison J, Short WR, Yawetz S, Ciaranello A, Livingston E, Duthely L, Rimawi BH, Anderson JR, Stringer EM; HOPES (HIV OB Pregnancy Education Study) Group. Integrase inhibitors in late pregnancy and rapid HIV viral load reduction. Am J Obstet Gynecol. 2016 Mar;214(3):385.e1-7. doi: 10.1016/j.ajog.2015.12.052. PMID 26928154
- [Background] Rutherford GW, Horvath H. Dolutegravir Plus Two Nucleoside Reverse Transcriptase Inhibitors versus Efavirenz Plus Two Nucleoside Reverse Transcriptase Inhibitors As Initial Antiretroviral Therapy for People with HIV: A Systematic Review. PLoS One. 2016 Oct 13;11(10):e0162775. doi: 10.1371/journal.pone.0162775. eCollection 2016. PMID 27736859
- [Background] Phillips AN, Stover J, Cambiano V, Nakagawa F, Jordan MR, Pillay D, Doherty M, Revill P, Bertagnolio S. Impact of HIV Drug Resistance on HIV/AIDS-Associated Mortality, New Infections, and Antiretroviral Therapy Program Costs in Sub-Saharan Africa. J Infect Dis. 2017 May 1;215(9):1362-1365. doi: 10.1093/infdis/jix089. PMID 28329236
- [Background] Van Laethem K, Schrooten Y, Covens K, Dekeersmaeker N, De Munter P, Van Wijngaerden E, Van Ranst M, Vandamme AM. A genotypic assay for the amplification and sequencing of integrase from diverse HIV-1 group M subtypes. J Virol Methods. 2008 Nov;153(2):176-81. doi: 10.1016/j.jviromet.2008.07.008. Epub 2008 Sep 2. PMID 18706932
- [Background] Van Zyl GU, Liu TF, Claassen M, Engelbrecht S, de Oliveira T, Preiser W, Wood NT, Travers S, Shafer RW. Trends in Genotypic HIV-1 Antiretroviral Resistance between 2006 and 2012 in South African Patients Receiving First- and Second-Line Antiretroviral Treatment Regimens. PLoS One. 2013 Jun 26;8(6):e67188. doi: 10.1371/journal.pone.0067188. Print 2013. PMID 23840622
- [Derived] van Zyl GU, Decloedt E, Jennings L, Kellermann T, Motha K, van Schalkwyk M, Schreuder C, Coetzee N, Glidden DV, Orrell C, Gandhi M. A Real-Time Urine Tenofovir Assay Improves Drug Adherence Among People With HIV With Prior Virologic Failure in a Randomized Controlled Trial. Clin Infect Dis. 2025 Dec 24;81(5):e352-e359. doi: 10.1093/cid/ciaf337. PMID 40578842

DOCUMENTS (2):
  • Study Protocol (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT05333679/Prot_000.pdf
  • Informed Consent Form (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/79/NCT05333679/ICF_002.pdf